CLINICAL TRIAL: NCT00315367
Title: A Double-Blind, Crossover Trial of Aricept® in Memory-Impaired Patients With Multiple Sclerosis: A Phase IV Demonstration of Functional MRI (fMRI) as a Surrogate Marker of Brain Activity Associated With Improvement in Memory Function
Brief Title: A fMRI(Functional Magnetic Resonance Imaging) Research Study to Learn More About Multiple Sclerosis and Individuals Potentially Experiencing Memory Difficulties
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neurognostics (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MSA1-904
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2007-10-16 (Estimated); Status verified 2007-10

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Memory impairment
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Memory Disorders | interventions — Pharmaceutical Preparations

INTERVENTIONS:
Drug: Donepezil HCI (drug)

SUMMARY:
The purpose of this study is to determine if medication designed to improve memory will help patients with Multiple Sclerosis (MS) who are experiencing memory problems using fMRI to track brain activity.

DETAILED DESCRIPTION:
Donepezil HCI (Aricept®) is an FDA-approved drug now used to enhance memory in patients with Alzheimer's disease. The aim of this project is to examine the effects of Donepezil HCI (Aricept®) on memory induced brain activation patterns in the context of a double-blind, crossover trial of patients with multiple sclerosis (MS). We will perform task activation experiments involving two cognitive domains. The proposed work on MS patients should yield new information regarding functional anatomic relationships during cognitive activity, and how these relationships change as a function of drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age and experiencing some forgetfulness
* Diagnosed with MS, currently taking Rebif® and experiencing mild memory problems
* Participants will have stable medication dosages 1 month prior to testing
* With no past or present neurological disorders (e.g. head trauma, seizures, encephalitis, stroke) except MS
* With no known medical illnesses (e.g. diabetes, uncontrolled hypertension, arthritis)
* With no psychiatric illness
* With no current substance abuse
* Females should not be pregnant or nursing
* With no metallic devices in the body or claustrophobia

Exclusion Criteria:

* Previous history of CNS disturbance other than MS
* Severe motor or visual impairment that might interfere with the cognitive activation tasks
* Prescribed psychoactive medications
* Memory deficits caused by other significant neurological disease or psychiatric disorder
* Active malignancy within one year of study participation
* Known human immunodeficiency virus (HIV)
* Current diagnosis of unstable glaucoma; history of myocardial infarction
* Symptomatic Coronary Artery Disease within the last 12 months or evidence of ongoing ischemia or uncontrolled atrial or ventricular arrhythmias as shown by ECG; poorly controlled or labile hypertension
* History of epilepsy or other seizure disorder within the past 12 months
* Allergy or hypersensitivity to amphetamines or other sympathomimetic amines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2004-09; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Anatomic relationships during cognitive activity, and how these relationships change as a function of drug

SECONDARY OUTCOMES:
fMRI as a surrogate marker for drug efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Safwan Jaradeh, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Krupp LB, Christodoulou C, Melville P, Scherl WF, MacAllister WS, Elkins LE. Donepezil improved memory in multiple sclerosis in a randomized clinical trial. Neurology. 2004 Nov 9;63(9):1579-85. doi: 10.1212/01.wnl.0000142989.09633.5a. PMID 15534239